CLINICAL TRIAL: NCT00290875
Title: Implementation of the Canadian C-Spine Rule: Phase III
Brief Title: Implementation of the Canadian C-Spine Rule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. I. Stiell, Senior Scientist, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2002174-01H, MOP62795; 2002174-01H
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Cspine Injury
Keywords: cspine injury; radiography; clinical impact; dissemination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): We randomly allocated sites to either intervention or control. At the intervention sites, active strategies were employed to implement the rule into practice, including education, policy, and real-time reminders on radiology requisitions.
  Interventions: Behavioral: Use of Xrays for diagnosis

INTERVENTIONS:
Behavioral: Use of Xrays for diagnosis

SUMMARY:
Many thousands of trauma patients are seen in Canadian emergency departments each year. On rare occasions, such patients have a broken neck (cervical spine fracture) but in 98 percent of cases the xrays ordered by the doctors are normal. The total cost of inexpensive but high volume tests such as neck x-rays adds considerably to rising health care costs. In addition, these patients are often immobilized with uncomfortable backboards and collars for many hours, tying up valuable space and time in our crowded emergency departments.

This research group recently developed and tested a highly accurate and reliable guideline called the Canadian C-Spine Rule to help physicians be much more selective in their use of neck x-rays and to minimize the period of immobilization. This research project will evaluate the true effectiveness of the Rule when implemented with simple and inexpensive measures. This study will involve 14,000 patients in 12 busy emergency departments across Canada.

This Canadian C-Spine Rule is designed to allow physicians to be much more selective in their use of neck xrays without the risk of missing a fracture or dislocation of the neck and to reduce the length of time of immobilization. Widespread use of the guideline could lead to large savings for our health care systems without jeopardizing patients and could greatly expedite care of trauma patients in our crowded emergency departments.

DETAILED DESCRIPTION:
Background: Physicians in Canadian emergency departments (EDs) annually treat 185,000 alert and stable trauma victims who are at risk for cervical spine (c-spine) injury. Only 0.9% of these patients have, however, suffered a cervical spine fracture. Current use of radiography is not efficient. More than 98% of c-spine radiographs are negative and there is considerable variation among hospitals and physicians in radiography use. C-spine radiographs are little ticket items, low cost procedures that significantly add to health care costs due to high volume. In addition, alert and stable trauma patients are often immobilized on a backboard with a rigid collar and sandbags for many hours. This leads to considerable patient discomfort and unnecessary use of valuable time and space in our crowded EDs. This renewal application builds on previous MRC/CIHR grants to determine feasibility (phase 0, MRC GR-13304D, 1995-96), develop a decision rule for c-spine radiography (phase I, MRC MT-13700, 1996-99, N=8,924), and prospectively validate this Canadian C-Spine Rule (phase II, CIHR MT13700, 1999-2002, N=8,000), all part of the University of Ottawa Group Grant in Decision Support Techniques (CIHR 2000-143). The Canadian C-Spine Rule is comprised of simple clinical variables (Figure 1) and allows physicians to be much more selective in ordering radiography (JAMA 2001). In the recently completed prospective validation (phase II), we confirmed the accuracy and reliability of the rule.

Objectives: The goal of phase III is to evaluate the effectiveness and safety of an active strategy to implement the Canadian C-Spine Rule into physician practice. Specific objectives are to: 1) Determine clinical impact by comparing the intervention and control sites for: a) C-spine radiography rates, b) Missed fractures, c) Serious adverse outcomes, d) Length of stay in ED, and e) Patient satisfaction; 2) Determine sustainability of the impact; 3) Evaluate performance of the Canadian C-Spine Rule, with regards to: a) Accuracy, b) Physician accuracy in interpretation, and c) Physician comfort and compliance with use; 4) Conduct an economic evaluation to determine the potential for cost savings with widespread implementation.

Methods: We propose a matched-pair cluster design study which compares outcomes during 3 consecutive 12-month before, after, and decay periods at 6 pairs of intervention and control sites (Figure 3). These 12 hospital ED sites will be stratified as teaching or community hospitals, matched according to baseline c-spine radiography ordering rates, and then allocated within each pair to either intervention or control groups. During the after period at the intervention sites, simple and inexpensive strategies will be employed to actively implement the Canadian C-Spine Rule: a) physician group discussion and consensus, b) educational initiatives (lecture, posters, pocket cards), and c) a process-of-care modification with a mandatory reminder of the Rule at the point of requisition for radiography. These outcomes will be assessed: 1) Measures of clinical impact will compare the changes from before to after between the intervention and control sites: a) C-spine radiography ordering proportions (the primary analysis); b) Number of missed fractures; c) Number of serious adverse outcomes; d) Length of stay in ED; e) Patient satisfaction. 2) Performance of the Canadian C-Spine Rule: a) Accuracy of the rule; b) Physician accuracy of interpretation; c) Physician comfort and compliance. 3) Economic evaluation measures: a) Radiography rate after discharge; b) Length of stay in ED and hospital; c) Hospital admission; d) Operative repair. During the 12-month decay period, implementation strategies will continue, allowing us to evaluate the sustainability of the effect. We estimate a sample size of 4,800 patients in each period in order to have adequate power to evaluate the main outcomes.

Importance: This implementation study (phase III) is an essential step in the process of developing a new clinical decision rule guideline for health care practitioners. Phase I successfully derived the Canadian C-Spine Rule and phase II confirmed the accuracy and safety of the rule and, hence, the potential for physicians to improve care. What remains unknown is the actual change in clinical behaviour that can be effected by implementation of the Canadian C-Spine Rule and whether implementation can be achieved with simple and inexpensive measures. We believe that the Canadian C-Spine Rule has the potential to significantly reduce health care costs and improve the efficiency of patient flow in busy Canadian EDs.

ELIGIBILITY:
Inclusion Criteria:All alert, stable adults presenting to the study hospital EDs after sustaining acute blunt trauma to the head or neck will be eligible and consecutive eligible trauma patients will be entered into the study. Patient eligibility will be determined based on these criteria at the time of arrival in the ED. a) "Trauma to the head and neck" will include patients with either: i) neck pain with any mechanism of injury (subjective complaint by the patient of any pain in the posterior midline or posterolateral aspect of the neck), or ii) no neck pain but all of: some visible injury above the clavicles, has not been ambulatory at any time, and associated with a high risk mechanism of injury (motor vehicle collision including motorcycle, pedestrian struck by a motor vehicle, bicycle collision, fall greater than or equal to 3 feet or 5 steps, diving, or contact sport with axial load to head and neck). b) "Alert" is defined as a Glasgow Coma Scale103 score of 15 (converses, fully oriented, and follows commands). c) "Stable" refers to normal vital signs as defined by the Revised Trauma Score24 (systolic blood pressure 90 mm Hg or greater and respiratory rate between 10 and 24 breaths per minute). d) "Acute" refers to injury within the past 48 hours.

-

Exclusion Criteria:a) Patients under the age of 16 years, b) Patients who do not satisfy the definition of "trauma to the head and neck" as defined above (for example, patients with neither neck pain nor visible injuries above the clavicles will be excluded), c) Patients with Glasgow Coma Scale score less than 15, d) Patients with unstable vital signs (systolic BP < 90; respiratory rate less than 10 or more than 24), e) Patients whose injury occurred more than 48 hours previously, f) Patients with penetrating trauma from stabbing or gunshot wound, g) Patients with acute paralysis (paraplegia, quadriplegia), h) Patients with known vertebral disease (ankylosing spondylitis, rheumatoid arthritis, spinal stenosis, or previous cervical spine surgery), or i) Patients who return for reassessment of the same injury.

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11824 (Actual)
Dates: Start 2003-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Cervical spine radiography ordering proportions | 12 months
  The primary study outcome was the proportion of eligible patients referred for diagnostic imaging of the cervical spine. Daily patient census logs were reviewed to identify potential injury patients and patient eligibility was determined from emergency department nursing and physician records and ambulance reports. Radiology reports and census lists were reviewed to determine if cervical spine imaging was performed.

SECONDARY OUTCOMES:
Number of missed CSI Number of serious adverse outcomes Length of stay in ED Patient satisfaction Sustainability of the intervention Performance of the Canadian C-Spine Rule Economic evaluation measures | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ian Stiell, MD, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Stiell IG, Clement CM, Grimshaw J, Brison RJ, Rowe BH, Schull MJ, Lee JS, Brehaut J, McKnight RD, Eisenhauer MA, Dreyer J, Letovsky E, Rutledge T, MacPhail I, Ross S, Shah A, Perry JJ, Holroyd BR, Ip U, Lesiuk H, Wells GA. Implementation of the Canadian C-Spine Rule: prospective 12 centre cluster randomised trial. BMJ. 2009 Oct 29;339:b4146. doi: 10.1136/bmj.b4146. PMID 19875425